CLINICAL TRIAL: NCT04004143
Title: Micronutrients and Health in Adult Chinese
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Chronic Disease Control (Other)
Collaborators: Sun Yat-sen University (Other); Shenzhen Qilinshan Sanatorium (Unknown)
Responsible Party: Principal Investigator, Zhou Ji-Chang, Principal Investigator, Shenzhen Center for Chronic Disease Control
Other Study IDs: QLS2014
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Dysglycemia; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples were collected and separated by centrifugation for supernatant and blood cells.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-sectional: a cross-sectional study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
Adult subjects were recruited from a health examination center. Their fasting blood samples were collected for laboratory analyses of multiple measures including mineral, glucose, lipids, etc.

ELIGIBILITY:
Inclusion Criteria:

* adult volunteer
* Han population
* living in Shenzhen City for > 2 y

Exclusion Criteria:

* caught by organic diseases
* in pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers visiting a health examination center were randomly recruited with their consent to particiapate the study.
Sampling Method: Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
circulation concentration of glucose | less than 4 hours
  Glucose (mmol/L) was measured in less than 4 hours after sample collection
circulation concentrations of 4 types of lipids | less than 4 hours
  TG, TC, LDLC, and HDLC (mmol/L) were measured in less than 4 hours after sample collection
circulation concentrations of 5 minerals | less than 3 years
  all samples were stored at minus 75 degrees Celsius until ready for analysis collectively on a ICP-MS machine for calcium, cobalt, iron, selenium, and zinc (ng/ml)

SECONDARY OUTCOMES:
body mass index | less than 1 month
  body weight (kg) and hight (m) were measured when the volunteers were visiting the health examination center, and the body mass index was calculated later by the formula of body weight/ hight/ hight (kg/m^2).
circulation concentration of 25OHD | less than 3 years
  all samples were stored at minus 75 degrees Celsius until ready for analysis collectively with ELISA kits (nmol/L)